CLINICAL TRIAL: NCT00653185
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate Weekly Treatment With SYR-472 in Subjects With Type 2 Diabetes
Brief Title: Efficacy of SYR-472 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-SYR-472-007; U1111-1183-0302 (Registry Identifier: WHO)
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias; Hyperglycemia | interventions — trelagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- SYR-472 25 mg QD (Experimental): (with lifestyle modification and/or metformin therapy)
  Interventions: Drug: SYR-472
- SYR-472 50 mg QD (Experimental): (with lifestyle modification and/or metformin therapy)
  Interventions: Drug: SYR-472
- SYR-472 100 mg QD (Experimental): (with lifestyle modification and/or metformin therapy)
  Interventions: Drug: SYR-472
- SYR-472 200 mg QD (Experimental): (with lifestyle modification and/or metformin therapy)
  Interventions: Drug: SYR-472
- Placebo QD (Placebo Comparator): (with lifestyle modification and/or metformin therapy)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYR-472 — SYR-472 25 mg, tablets, orally, once daily and lifestyle modification and/or metformin for up to 12 weeks.
  Arms: SYR-472 25 mg QD
Drug: SYR-472 — SYR-472 50 mg, tablets, orally, once daily and lifestyle modification and/or metformin for up to 12 weeks.
  Arms: SYR-472 50 mg QD
Drug: SYR-472 — SYR-472 100 mg, tablets, orally, once daily and lifestyle modification and/or metformin for up to 12 weeks.
  Arms: SYR-472 100 mg QD
Drug: SYR-472 — SYR-472 200 mg, tablets, orally, once daily and lifestyle modification and/or metformin for up to 12 weeks.
  Arms: SYR-472 200 mg QD
Drug: Placebo — SYR-472 placebo-matching tablets, orally, once daily and lifestyle modification and/or metformin for up to 12 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the efficacy, safety and tolerability of SYR-472, once daily (QD), in subjects with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a complex metabolic disorder characterized by abnormal insulin secretion and glucose homeostasis, resulting from impaired pancreatic beta-cell function and insulin resistance in target tissues. The worldwide prevalence of type 2 diabetes mellitus is reaching epidemic proportions, and the total number of cases is expected to reach 221 million by 2010. The high incidence of the disease and its associated complications places a significant burden on healthcare systems.

The primary risk factor for the development of type 2 diabetes mellitus is obesity and its associated insulin resistance. Insulin resistance is characterized by an impaired response to the physiologic effects of insulin and leads to decreased cellular glucose uptake, increased hepatic gluconeogenesis, and a compensatory increase in insulin secretion that contributes to beta-cell exhaustion. Therefore in the insulin-resistant state, blood glucose and insulin levels are increased. The relationship between improved glycemic control in patients with type 2 diabetes mellitus and the delay or prevention of comorbidities has been reported in the Diabetes Control and Complications Trial and the United Kingdom Prospective Diabetes Study. Therefore, reduction of persistent hyperglycemia is the highest priority in treating this disease.

Diet and exercise are important and effective measures for maintaining glycemic control in individuals with insulin resistance, impaired glucose tolerance, and type 2 diabetes mellitus, particularly in the early stages of disease progression. In cases where diet and exercise alone fail to adequately maintain glycemic control, oral antidiabetic drugs are typically used. Combination oral therapy and eventually insulin are usually required to maintain lower blood glucose levels but can result in adverse effects including hypoglycemia and weight gain. Therefore, novel safe and effective antidiabetic therapies are needed.

Dipeptidyl peptidase-4 is a ubiquitous aminopeptidase that is widely expressed in many tissues; it is thought to be primarily responsible for the in vivo degradation of at least two gut-derived incretin hormones, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide, which are both released in response to nutrient ingestion. Glucagon-like peptide-1 has been demonstrated to augment glucose-dependent insulin secretion; suppress glucagon release and hepatic gluconeogenesis; inhibit gastric emptying, and reduce appetite and food intake. Glucagon-like peptide-1 and glucose-dependent insulinotropic peptide also have been shown to promote insulin biosynthesis and stimulate beta cell proliferation and survival. Orally available inhibitors of dipeptidyl peptidase-4 activity have been developed that increase intact postprandial glucagon-like peptide-1 levels after oral administration.

SYR-472 is a selective inhibitor of dipeptidyl peptidase-4 in development to improve glycemic control in patients with type 2 diabetes mellitus. The aim of this study is to evaluate SYR-472 in subjects with type 2 diabetes mellitus who have not previously achieved adequate glycemic control with lifestyle modification (diet/exercise) or metformin antidiabetic monotherapy. Study participation is anticipated to be up to 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a historical diagnosis of type 2 diabetes mellitus.
* Has undergone less than 7 days of any antidiabetic therapy except lifestyle modification (diet/exercise) within 8 weeks prior to Screening; or has received metformin monotherapy for at least 8 weeks prior to Screening and maintained a stable daily dose of metformin for at least 12 weeks prior to randomization.
* The subject receiving metformin monotherapy at randomization must have been at least 75% compliant with his or her regimen during the Run-in/Stabilization Period as determined by subject diary and investigator assessment.
* Has received no treatment with antidiabetic agents other than metformin within the 8 weeks prior to Screening.
* Has a glycosylated hemoglobin concentration between 7.0% and 10.0%, inclusive, at Screening and at the Week -1 Visit.
* The subject's fasting C-peptide concentration is greater than or equal to 0.8 ng/mL.
* Has a fasting plasma glucose concentration less than 275 mg/dL.
* If regularly uses other non-excluded medications, must be on a stable dose for at least the 4 weeks prior to Screening.
* Has a systolic blood pressure reading less than 160 mm Hg and a diastolic pressure reading less than 100 mm Hg.
* Has a hemoglobin value greater than or equal to 12 g/dL for men and greater than or equal to 10 g/dL for women.
* Has an alanine aminotransferase level is less than or equal to 3 times the upper limit of normal.
* Males have a serum creatinine value less than 1.5 mg/dL; females have a serum creatinine value less than 1.4 mg/dL.
* Has a urine albumin/creatinine ratio less than 1000 μg/mg.
* Has a thyroid-stimulating hormone level less than or equal to the upper limit of the normal range and is clinically euthyroid.
* Females must be not be pregnant or lactating, and must agree to use adequate contraception throughout the duration of the study.
* Is able and willing to monitor his or her own blood glucose concentrations with a home glucose monitor.
* Has no major illness or debility that in the investigator's opinion prohibits the subject from completing the study.

Exclusion Criteria

* Is being concurrently treated with antidiabetic therapy other than metformin and lifestyle intervention.
* Has a history of cancer, other than squamous cell or basal cell carcinoma of the skin that has not been in full remission for at least 5 years prior to Screening.
* Has a history of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* Has a history of treated diabetic gastric paresis.
* Has New York Heart Association class III or IV heart failure regardless of therapy.
* Has a history of coronary angioplasty, underwent coronary stent placement or coronary bypass surgery, or suffered a myocardial infarction, or stroke within the 6 months prior to Screening.
* Has a history of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* Has a history of infection with human immunodeficiency virus.
* Has a history of a psychiatric disorder that in the investigator's opinion will affect the subject's ability to participate in the study.
* Has ingested or received systemically injected glucocorticoids within the 3 months prior to randomization. Inhaled corticosteroids are allowed.
* Has used prescription or over-the-counter weight-loss drugs within the 3 months prior to randomization.
* Has received any investigational drug within the 30 days prior to Screening or has received an investigational antidiabetic drug within the 3 months prior to Screening.
* Has received previous treatment in an investigational study of SYR-472.
* Has a known hypersensitivity to any compound related to SYR-472.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin | Weeks 12 or Final Visit.

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin | Weeks 4, 8, and 12 or Final Visit.
Change from baseline in fasting plasma glucose | Weeks 1, 2, 4, 8, and 12 or Final Visit.
1,5-Anhydroglucitol | Weeks 2, 4, 8, and 12 or Final Visit.
Change in Proinsulin | Weeks 4, 8, and 12 or Final Visit.
Change in Proinsulin/insulin ratio | Weeks 4, 8, and 12 or Final Visit.
Change in baseline C-peptide | Weeks 4, 8, and 12 or Final Visit.
Change from baseline in insulin | Weeks 4, 8, and 12 or Final Visit.
Change in Homeostasis model assessment of beta cell function | Weeks 4, 8, and 12 or Final Visit.
Change in Homeostasis model assessment of insulin resistance | Weeks 4, 8, and 12 or Final Visit
Incidence of rescue | Weeks 1, 2, 4, 8, and 12 or Final Visit.
Clinical response endpoint incidence of glycosylated hemoglobin less than or equal to 6.5% | Week 12 or Final Visit
Clinical response endpoint incidence of glycosylated hemoglobin less than or equal to 7.0% | Week 12 or Final Visit
Change from baseline in Fasting lipids (triglycerides, total cholesterol, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol) | Weeks 4, 8, and 12 or Final Visit
Body weight | Weeks 4, 8, and 12 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (87):
- United States (51):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Pell City, Alabama
  - Tallassee, Alabama
  - Sierra Vista, Arizona
  - Fountain Valley, California
  - Los Angeles, California
  - National City, California
  - Pismo Beach, California
  - Clearwater, Florida
  - North Miami Beach, Florida
  - Ocoee, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Dawsonville, Georgia
  - Gainesville, Georgia
  - Naperville, Illinois
  - Elkhart, Indiana
  - Indianapolis, Indiana
  - Slidell, Louisiana
  - Taunton, Massachusetts
  - Ann Arbor, Michigan
  - Great Falls, Montana
  - Scottsbluff, Nebraska
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Charlotte, North Carolina
  - Shelby, North Carolina
  - Sparta, North Carolina
  - Fargo, North Dakota
  - Bensalem, Ohio
  - Dayton, Ohio
  - Kettering, Ohio
  - Central Point, Oregon
  - Altoona, Pennsylvania
  - Providence, Rhode Island
  - Clemson, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Rapid City, South Dakota
  - Cleveland, Tennessee
  - Kingsport, Tennessee
  - Arlington, Texas
  - Fort Worth, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Sugarland, Texas
  - Hampton, Virginia
  - Richmond, Virginia
- Chile (2):
  - Santiago
  - Temuco
- Czechia (2):
  - Ostrava
  - Prague
- Guatemala (2):
  - Guatemala City
  - Quetzaltenango
- Hungary (2):
  - Eger
  - Szentes
- Latvia (3):
  - Riga
  - Sigulda
  - Valmiera
- Lithuania (4):
  - Kaunas
  - Kėdainiai
  - Klaipėda
  - Vilnius
- Ponce, Puerto Rico
- Romania (9):
  - Alba Iulia
  - Baia Mare
  - Bihor
  - Brasov
  - Bucharest
  - Constanța
  - Ploieşti
  - Satu Mare
  - Târgovişte
- Russia (6):
  - Kemerovo
  - Moscow
  - Saint Petersburg
  - Ufa
  - Volgograd
  - Yaroslavl
- Slovakia (3):
  - Banská Bystrica
  - Bratislava
  - Prešov
- Ukraine (2):
  - Kharkiv
  - Vinnytsia